CLINICAL TRIAL: NCT03897686
Title: Multicenter Double-blind Randomized Comparative Placebo-controlled Study of Efficacy and Safety of Intra-articular HBISA Endoprosthesis of Synovial Fluid (NOLTREX™) in Knee Osteoarthritis
Brief Title: Intra-articular Polyacrylamide Hydrogel in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Centre BIOFORM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA/PAAG-SI/OA/2019
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis
Keywords: intra-articular; polyacrylamide hydrogel; PAAG; Hydrous biopolymer with silver ions "Argiform" (HBISA); NOLTREX
MeSH Terms: conditions — Osteoarthritis | interventions — Abortion, Induced

STUDY DESIGN:
Intervention Model Description: multicenter double-blind randomized comparative placebo-controlled
Who Masked: Participant, Investigator
Masking Description: A patient, study investigator and Sponsor representative (monitoring specialist) will not know to which group a patient is included. to preserve blinding of any patient and study team, an independent unblended physician is to be engaged, he/she will receive the product per randomization code and perform the procedure of intra-articular injection of the study MD and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOLTREX™, OA grade II-III (Experimental): 72 patients with gonarthrosis grade II-III were randomised to receive PAHG
  Interventions: Device: hydrous biopolymer with silver ions "Argiform"
- Placebo,OA grade II-III (Placebo Comparator): 72 patients with gonarthrosis grade II-III were randomised to receive saline solution
  Interventions: Device: saline solution

INTERVENTIONS:
Device: hydrous biopolymer with silver ions "Argiform" — 2 once-weekly intra-articular injections of NOLTREX™ 4.0 ml
  Other Names: polyacrylamide hydrogel with silver ions; Synovial fluid endoprosthesis NOLTREX™
  Arms: NOLTREX™, OA grade II-III
Device: saline solution — 2 once-weekly intra-articular injections of saline solution 4 ml
  Arms: Placebo,OA grade II-III

SUMMARY:
The aim of this double-blinded controlled study is to assess clinical efficacy and safety of intra-articular HBISA Endoprosthesis of Synovial Fluid (polyacrylamide hydrogel) in comparison with placebo (0.9% sodium chloride solution) in Kellgren Lawrence radiological grade II-III knee osteoarthritis

DETAILED DESCRIPTION:
Polyacrylamide hydrogel (hereinafter - PAAG) is intended for a symptomatic effect leading to decrease of joint pain intensity and improvement of functional joint characteristics. Therefore PAAG is regarded as symptom-modifying therapy for joint osteoarthritis (hereinafter - OA). The aim of this study was to estimate efficacy and safety of intra-articular injections of PAAG in comparison with saline solution. Men and women above 50 years with verified knee osteoarthritis in accordance with the American College of Rheumatology (ACR) criteria were randomly assigned to one of 2 groups (PAAG or saline solution). Each patient received to the target knee joint one injection of 4.0 ml either PAAG or placebo with one-week interval. Course - 2 injections. To avoid the joint overfilling with the dense, slowly resorbing material in patients with a good clinical result, the course of injections was to be stopped. Primary and secondary efficacy endpoints, and safety parameters were assessed at weeks 6, 13 and 25 visits .

ELIGIBILITY:
Inclusion Criteria:

* Men and women above 50 years;
* Verified knee osteoarthritis in accordance with the ACR (knee pain combined with one of the following signs: age above 50 years, knee crepitus or morning joint stiffness lasting for less than 30 minutes combined with radiologic signs of knee osteoarthritis);
* Kellgren Lawrence radiological grade II-III knee osteoarthritis with the predominant involvement of the medial tibiofemoral region of the knee joint;
* Joint space width (JSW) of the target knee joint at least 2.5 mm.

Exclusion Criteria:

1. History of any injury or surgical intervention on the target knee joint (except for diagnostic arthroscopy made not longer than 60 days at the study entry);
2. Severe degenerative changes in the target knee joint determined as the joint space narrowing less than 2 mm;
3. Varus or valgus deformation of the target knee joint;
4. Instability of the target knee joint;
5. Active inflammation of the target knee joint (edema, hyperemia, present effusion) at the study entry;
6. Microcrystalline arthropathies;
7. Systemic inflammatory disease (rheumatoid arthritis, systemic lupus erythematosus, etc.);
8. Seronegative spondyloarthritis and reactive arthritis;
9. Inflammatory diseases of the skin and soft tissues in the proposed injection site for the test MD or placebo in the target joint;
10. History of venous thrombosis and thromboembolia;
11. Coagulogram abnormalities (APTT, prothrombin time, prothrombin index, fibrinogen);
12. Inflammatory changes in the complete blood count (leukocytosis, increase of erythrocyte sedimentation rate [ESR]);
13. Platelet count abnormality (in accordance with the reference ranges of the local laboratory;
14. Increase of rheumatoid factor level;
15. Increase of uric acid level > 360 μmol/l;
16. Diabetes mellitus;
17. Hemophilia and other hemorrhagic diatheses, as well administration of anticoagulants and disaggregants;
18. Positive results of HIV, HBs-Ag, anti-HCV, RW tests;
19. Intra-articular injection to the target knee joint:

    * Noltrex - within 24 months prior patient's inclusion to the study;
    * hyaluronates - within 6 months prior patient's inclusion to the study;
    * glucocorticosteroids - within 1 month prior the study inclusion;
    * non-steroidal anti-inflammatory drugs (NSAID) - within 3 weeks prior patient's inclusion to the study.
20. Oral administration of non-steroidal anti-inflammatory drugs (NSAID) within 2 weeks prior the study inclusion;
21. Necessity of systemic glucocorticosteroids in any dosage form;
22. Paracetamol administration within 48 hours prior the study inclusion;
23. Pregnancy and lactation;
24. Hypersensitivity to components of the test MD or placebo;
25. Severe liver disorder determined as the increase of one of the values: ALT, AST, ALP, total bilirubin, GGTP more than 3 times the upper limit of normal;
26. Renal diseases with the glomerular filtration rate estimated per Cockraft-Gault formula less than 60 ml/min/1.73 m2 (III-V stage chronic renal disease [CRD]);
27. Clinically manifest hip osteoarthritis;
28. History of knee and coxofemoral endoprosthesis;
29. Acute infectious diseases or infectious aggravations of chronic diseases (respiratory infections) within one month prior the study inclusion;
30. Severe decompensated chronic or acute diseases and other conditions which, by the opinion of the study physician, may preclude the patient's participation in the study or affect the study results.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir V Popov, DSc, Principal Investigator — Non-budgetary HCF "Railway clinical hospital n.a. Semashko N.A. at Lublino, OJSC "Russian Railways"
Locations (4):
- Russia (4):
  - Non-budgetary healthcare facility "Railway clinical hospital n.a. Semashko N.A. at Lublino, OJSC "Russian Railways", Moscow
  - "Clinical Diagnostic Center "Ultramed", LLC, Omsk
  - Private Healthcare Facilty "Clinical hospital "RZHD-Medicina" of the city Saint-Petersburg, Saint Petersburg
  - State budgetary healthcare facility of Yaroslavl Region "Clinical hospital №3", Yaroslavl

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 patients were selected for the study, of which 144 were randomised at 4 study sites from November 2019 to November 2020.
Pre-assignment Details: 7 patients were classified as "screen failure" and 144 patients were randomized (1:1) to receive NOLTREX™ (n = 72) or placebo (n = 72).
Groups:
- NOLTREX™, OA Grade II-III: 72 patients with knee osteoarthritis grade II-III received 2 weekly intra-articular injections of PAAG (NOLTREX™) 4.0 ml at the week 1 and 2 study visits
- Placebo, ОА Grade II-III: Patients with osteoarthritis Grade II-III received 2 weekly intra-articular injections of the saline solution (placebo) at the week 1 and 2 study visits.
Period: Overall Study
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Started | 72 | 72
Completed | 70 | 70
Not Completed | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were described by treatment group in the ITT population (all randomized patients who received at least one dose of study intervention)
Groups:
- NOLTREX™, OA Grade II-III: Patients with osteoarthritis Grade II-III received 2 weekly injections of the PAHG hydrous biopolymer with silver ions "Argiform" 4.0 ml (NOLTREX™) at the week 1 and 2 study visits.
- Placebo, OA Grade II-III: Patients with osteoarthritis Grade II-III received 2 weekly injections of the saline solution (placebo) at the week 1 and 2 study visits.
- Total: Total of all reporting groups
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, OA Grade II-III | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 63.40 (7.26) | 62.15 (7.54) | 62.775 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 117
  Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasoid | 72 | 72 | 144
  Race: Mongoloid | 0 | 0 | 0
  Race: Negroid | 0 | 0 | 0
  Race: Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Russia: Clinical center 1 | 3 | 3 | 6
  Russia: Clinical center 2 | 19 | 19 | 38
  Russia: Clinical center 3 | 10 | 10 | 20
  Russia: Clinical center 4 | 40 | 40 | 80
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.75 (2.97) | 29.44 (4.35) | 29.095 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Change of the Total WOMAC Score (WOMAC-T)
Description: Mean change from baseline (week 1) to visit 5 (Week 25) in the total WOMAC score. Patients were asked to complete the questionnaire during the study visit 5. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-500 for Pain, 0-200 for Stiffness, and 0-1700 for Physical Function. Higher scores represent worse pain, stiffness, and functional limitations. A sum of the scores for all three subscales gives a total WOMAC score (0-2400), where 0 represents the best health status and 2400 the worst possible status. The higher the score, the poorer the function.
Time Frame: baseline (week 1), week 25
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- NOLTREX™, OA Grade II-III: Patients with osteoarthritis Grade II-III received 2 weekly intra-articular injections of PAAG (NOLTREX™) 4.0 ml at the week 1 and 2 study visits.
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
score on a scale
  ОА grade II: number analyzed (Participants) | 61 | 56
  ОА grade II | -624.12 [-693.94 to -554.30] | -444.82 [-517.41 to -372.22]
  ОА grade II-III | -605.61 [-685.22 to -526.01] | -426.31 [-501.66 to -350.96]
  ОА grade III: number analyzed (Participants) | 11 | 16
  ОА grade III | -587.11 [-710.70 to -463.52] | -407.81 [-524.27 to -291.35]
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; It was determined that 144 participants randomized into 2 groups (1:1) would have at least 80% power to detect an effect size of 0.25. Sample size was calculated based on analysis of covariance adjusted for baseline value with fixed factors of group assuming α = 0.05 and 10% discontinuation rate. The null hypothesis states that there is no difference between treatment groups in mean change from baseline to Week 25 in the total WOMAC score; Test type: Superiority — [Not specified]; p = 0.00030, ANCOVA — The threshold for statistical significance was p <0.05; Analysis of covariance (ANCOVA) adjusted for the baseline value with fixed factors of "treatment group" and "radiological stage"; LS-means difference = -179.30, 95% CI 2-sided [-274.96 to -83.65], Standard Error of Mean 48.38
Statistical Analysis 2: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; After the analysis of covariance were performed pairwise comparisons of NOLTREX and placebo groups for each stage of OA: 1) Group A (NOLTREX™) OA grade II versus Group B (Placebo) ОА grade II; Test type: Superiority — [Not specified]; p = 0.0017, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -179.30, 95% CI 2-sided [-305.11 to -53.50], Standard Error of Mean 48.38
Statistical Analysis 3: Comparison: Placebo, ОА Grade II-III; After the analysis of covariance were performed pairwise comparisons of NOLTREX and placebo groups for each stage of OA: 2) Group A (NOLTREX™) OA grade II versus Group A (NOLTREX™) ОА grade III; Test type: Superiority; p = 0.9324, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -37.01, 95% CI 2-sided [-197.83 to 123.82], Standard Error of Mean 61.85
Statistical Analysis 4: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; After the analysis of covariance were performed pairwise comparisons of NOLTREX and placebo groups for each stage of OA: 3) Group A (NOLTREX™) OA grade II versus Group B (Placebo) ОА grade III; Test type: Superiority; p = 0.0233, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -216.31, 95% CI 2-sided [-411.37 to -21.25], Standard Error of Mean 75.01
Statistical Analysis 5: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; After the analysis of covariance were performed pairwise comparisons of NOLTREX and placebo groups for each stage of OA: 4) Group A (NOLTREX™) OA grade III versus Group B (Placebo) ОА grade II; Test type: Superiority; p = 0.3082, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = 142.30, 95% CI 2-sided [-70.63 to 355.22], Standard Error of Mean 81.89
Statistical Analysis 6: Comparison: NOLTREX™, OA Grade II-III; After the analysis of covariance were performed pairwise comparisons of NOLTREX and placebo groups for each stage of OA: 5) versus Group B (Placebo) OA grade II versus Group B (Placebo) ОА grade III; Test type: Superiority; p = 0.9324, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; LS-means difference = -37.01, 95% CI 2-sided [-197.83 to 123.82], Standard Error of Mean 61.85
Statistical Analysis 7: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; After the analysis of covariance were performed pairwise comparisons of NOLTREX and placebo groups for each stage of OA: 6) Group A (NOLTREX™) OA grade III versus Group B (Placebo) ОА grade III; Test type: Superiority; p = 0.0017, Tukey's HSD — Difference between Least-square means was tested at a level of p <0.05 via Tukey's multiple comparison test; Slope = -179.30, 95% CI 2-sided [-305.11 to -53.50], Standard Error of Mean 48.38

2. Secondary Outcome: Change of the Total WOMAC Score (WOMAC-T)
Description: Mean change from baseline (week 1) to Week 13 in the total WOMAC score. Patients were asked to complete the questionnaire during the study visits 1, 3, 4, 5. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores represent worse pain, stiffness, and functional limitations. A sum of the scores for all three subscales gives a total WOMAC score (0-96), where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function.
Time Frame: baseline (week 1), week 13 (visit 4)
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- NOLTREX™, OA Grade II-III: Patients with osteoarthritis Grade II-III received 2 weekly intra-articular injections of the PAHG hydrous biopolymer with silver ions "Argiform" 4.0 ml (NOLTREX™) at the week 1 and 2 study visits.
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
score on a scale | -532.57 [-609.74 to -455.40] | -389.18 [-461.99 to -316.37]
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; It was determined that 144 participants randomized into 2 groups (1:1) would have at least 80% power to detect an effect size of 0.25. Sample size was calculated based on analysis of covariance adjusted for baseline value with fixed factors of group assuming α = 0.05 and 10% discontinuation rate; Test type: Superiority — [Not specified]; p = 0.00267, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; S-means difference = -143.39, 95% CI 2-sided [-236.09 to -50.69], Standard Error of Mean 46.88

3. Secondary Outcome: The Pain Subscale Score WOMAC-A Changes
Description: Mean change from baseline (week 1) to week 6 (visit 3), 13 (visit 4) and 25 (visit 5) in the WOMAC Pain score (WOMAC-A). The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a set of standardized questionnaires used by health professionals to evaluate pain, stiffness and physical functioning of the joints in patients with knee and/or hip osteoarthritis. The WOMAC Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS. The WOMAC pain scale consists of five items: (1) walking on flat ground; (2) going up or down stairs; (3) at night while in bed; (4) sitting or lying; and (5) standing upright. The scores for the Pain subscale are summed up, with a possible score range of 0-500. Higher scores represent worse pain. Patients were asked to complete the questionnaire during the study visits 1, 3, 4, 5.
Time Frame: baseline (week 1), week 6 (visit 3), 13 (visit 4) and 25 (visit 5)
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
score on a scale
  Week 6 | -68.55 [-84.26 to -52.84] | -55.32 [-70.09 to -40.55]
  Week 13 | -110.94 [-127.40 to -94.48] | -84.24 [-99.71 to -68.77]
  Week 25 | -130.95 [-147.88 to -114.03] | -96.99 [-113.09 to -80.89]
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in pain WOMAC score at visit 3 (week 6); Test type: Superiority; p = 0.16786, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -13.23, 95% CI 2-sided [-32.096 to 5.638], Standard Error of Mean 9.995
Statistical Analysis 2: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in pain WOMAC score at visit 4 (week 13); Test type: Superiority; p = 0.00847, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -26.695, 95% CI 2-sided [-46.46 to -6.93], Standard Error of Mean 9.995
Statistical Analysis 3: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in pain WOMAC score at visit 5 (week 25); Test type: Superiority; p = 0.00123, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -33.96, 95% CI 2-sided [-54.31 to -13.62], Standard Error of Mean 10.29

4. Secondary Outcome: The Stiffness (WOMAC-B) and Functionality (WOMAC-C) Subscale Scores Changes
Description: Mean change from baseline (week 1) to week 6 (visit 3), 13 (visit 4) and 25 (visit 5) in the WOMAC Stiffness (WOMAC-B) and WOMAC Physical Function (WOMAC-C) scores. Patients were asked to complete the questionnaire during the study visit 5. The Western Ontario and McMaster Universities Osteoarthritis Index Version 3.1 Visual Analog Scale Format (WOMAC VA 3.1) applies a 100 mm VAS and consists of three subscales: pain (5 questions), stiffness (2 questions), and physical function (17 questions). The scores for each subscale are summed up, with a possible score range of 0-200 for Stiffness, and 0-1700 for Physical Function. Higher scores represent worse stiffness and functional limitations. The higher the score, the poorer the function.
Time Frame: baseline (week 1), week 6 (visit 3), 13 (visit 4) and 25 (visit 5)
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
score on a scale
  WOMAC-B /Week 6 | -27.25 [-35.68 to -18.81] | -27.10 [-35.06 to -19.14]
  WOMAC-B /Week 13 | -48.46 [-57.16 to -39.74] | -33.96 [-42.18 to -25.74]
  WOMAC-B /Week 25 | -54.79 [-62.48 to -47.10] | -38.61 [-45.96 to -31.25]
  WOMAC-C /Week 6 | -240.41 [-293.24 to -187.58] | -183.26 [-233.13 to -133.39]
  WOMAC-C /Week 13 | -374.17 [-430.00 to -318.34] | -270.90 [-323.60 to -218.20]
  WOMAC-C /Week 25 | -436.92 [-494.86 to -378.97] | -303.63 [-359.00 to -248.26]
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in stiffness WOMAC score, visit 3; Test type: Superiority; p = 0.97733, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -0.146, 95% CI 2-sided [-10.271 to 9.980], Standard Error of Mean 5.121
Statistical Analysis 2: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in stiffness WOMAC score, visit 4; Test type: Superiority; p = 0.00693, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -14.50, 95% CI 2-sided [-24.95 to -4.04], Standard Error of Mean 5.29
Statistical Analysis 3: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in pain WOMAC score at visit 5 (week 25); Test type: Superiority; p = 0.00073, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -16.18, 95% CI 2-sided [-25.44 to -6.92], Standard Error of Mean 4.68
Statistical Analysis 4: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in functionality WOMAC score, visit 3; Test type: Superiority; p = 0.07725, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -57.14, 95% CI 2-sided [-120.62 to 6.33], Standard Error of Mean 32.10
Statistical Analysis 5: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in functionality WOMAC score, visit 4; Test type: Superiority; p = 0.00279, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -103.27, 95% CI 2-sided [-170.35 to -36.20], Standard Error of Mean 33.92
Statistical Analysis 6: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; Contrasts for changes in functionality WOMAC score, visit 5; Test type: Superiority; p = 0.00023, ANCOVA — The threshold for statistical significance was p <0.05; [statistical method as in outcome 1, analysis 1]; LS-means difference = -133.29, 95% CI 2-sided [-203.03 to -63.55], Standard Error of Mean 35.26

5. Secondary Outcome: Patient Assessment of Treatment Efficacy
Description: Patient satisfaction with treatment was measured by a 6-point scale Likert scale (evident aggravation, aggravation, without changes, weak improvement, improvement, significant improvement) at the study visits 3 (week 6), 4 (week 13) and 5 (week 25).
Time Frame: Week 6, Week 13 and Week 25
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- PlLACEBO, ОА Grade II-III: Patients with osteoarthritis Grade II-III received 2 weekly intra-articular injections of the saline solution (placebo) at the week 1 and 2 study visits.
Arm/Group | NOLTREX™, OA Grade II-III | PlLACEBO, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
participants
  Week 6, evident aggravation: number analyzed (Participants) | 71 | 72
  Week 6, evident aggravation | 0 [0.00 to 13.49] | 0 [0.00 to 13.33]
  Week 6,aggravation: number analyzed (Participants) | 71 | 72
  Week 6,aggravation | 0 [0.00 to 13.49] | 4 [1.23 to 21.73]
  Week 6, without changes: number analyzed (Participants) | 71 | 72
  Week 6, without changes | 17 [11.40 to 43.52] | 21 [15.12 to 48.77]
  Week 6, weak improvement: number analyzed (Participants) | 71 | 72
  Week 6, weak improvement | 18 [12.36 to 45.00] | 30 [24.75 to 60.81]
  Week 6, improvement: number analyzed (Participants) | 71 | 72
  Week 6, improvement | 27 [21.74 to 57.55] | 13 [7.64 to 36.99]
  Week 6, significant improvement: number analyzed (Participants) | 71 | 72
  Week 6, significant improvement | 9 [4.49 to 30.93] | 4 [1.23 to 21.73]
  Week 13,evident aggravation: number analyzed (Participants) | 71 | 72
  Week 13,evident aggravation | 0 [0.00 to 13.49] | 0 [0.00 to 13.33]
  Week 13,aggravation: number analyzed (Participants) | 71 | 72
  Week 13,aggravation | 0 [0.00 to 13.49] | 4 [1.23 to 21.73]
  Week 13, without changes: number analyzed (Participants) | 71 | 72
  Week 13, without changes | 5 [1.80 to 23.88] | 17 [11.23 to 43.03]
  Week 13, weak improvement: number analyzed (Participants) | 71 | 72
  Week 13, weak improvement | 18 [12.36 to 45.00] | 25 [19.26 to 54.26]
  Week 13, improvement: number analyzed (Participants) | 71 | 72
  Week 13, improvement | 33 [28.63 to 65.28] | 19 [13.14 to 45.93]
  Week 13, significant improvement: number analyzed (Participants) | 71 | 72
  Week 13, significant improvement | 15 [9.53 to 40.51] | 7 [3.02 to 27.16]
  Week 25,evident aggravation: number analyzed (Participants) | 70 | 70
  Week 25,evident aggravation | 0 [0.00 to 13.66] | 0 [0.00 to 13.66]
  Week 25, aggravation: number analyzed (Participants) | 70 | 70
  Week 25, aggravation | 0 [0.00 to 13.66] | 2 [0.39 to 18.20]
  Week 25, without changes: number analyzed (Participants) | 70 | 70
  Week 25, without changes | 6 [2.44 to 26.02] | 19 [13.54 to 46.99]
  Week 25, weak improvement: number analyzed (Participants) | 70 | 70
  Week 25, weak improvement | 14 [8.76 to 39.44] | 20 [14.55 to 48.45]
  Week 25, improvement: number analyzed (Participants) | 70 | 70
  Week 25, improvement | 30 [25.52 to 62.15] | 20 [14.55 to 48.45]
  Week 25, significant improvement: number analyzed (Participants) | 70 | 70
  Week 25, significant improvement | 20 [14.55 to 48.45] | 9 [4.56 to 31.30]
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs PlLACEBO, ОА Grade II-III; The Chi-Square test was used to determine whether there was a statistically significant difference in disposition of results between two groups; Test type: Superiority; p < 0.005, Chi-squared — The level of significance was set to p <0.05; P-value generated by Chi-squared test was ≤0.005 for each time point

6. Secondary Outcome: Investigator Assessment of Treatment Efficacy
Description: Investigator satisfaction with treatment was measured by a 6-point scale Likert scale (evident aggravation, aggravation, without changes, weak improvement, improvement, significant improvement) at the study visits 3 (week 6), 4 (week 13) and 5 (week 25).
Time Frame: Week 6, Week 13 and Week 25
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | NOLTREX™, OA Grade II-III | PLACEBO, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
participants
  Week 6, evident aggravation: number analyzed (Participants) | 71 | 72
  Week 6, evident aggravation | 0 [0.00 to 13.49] | 0 [0.00 to 13.33]
  Week 6,aggravation: number analyzed (Participants) | 71 | 72
  Week 6,aggravation | 0 [0.00 to 13.49] | 1 [0.11 to 15.63]
  Week 6, without changes: number analyzed (Participants) | 71 | 72
  Week 6, without changes | 17 [11.40 to 43.52] | 28 [22.51 to 58.23]
  Week 6, weak improvement: number analyzed (Participants) | 71 | 72
  Week 6, weak improvement | 18 [12.36 to 45.00] | 26 [20.33 to 55.59]
  Week 6, improvement: number analyzed (Participants) | 71 | 72
  Week 6, improvement | 28 [22.86 to 58.87] | 14 [8.51 to 38.53]
  Week 6, significant improvement: number analyzed (Participants) | 71 | 72
  Week 6, significant improvement | 8 [3.76 to 29.23] | 3 [0.76 to 19.79]
  Week 13,evident aggravation: number analyzed (Participants) | 71 | 72
  Week 13,evident aggravation | 0 [0.00 to 13.49] | 0 [0.00 to 13.33]
  Week 13,aggravation: number analyzed (Participants) | 71 | 72
  Week 13,aggravation | 0 [0.00 to 13.49] | 1 [0.11 to 15.63]
  Week 13, without changes | 7 [3.06 to 27.49] | 23 [17.16 to 51.54]
  Week 13, weak improvement: number analyzed (Participants) | 71 | 72
  Week 13, weak improvement | 18 [12.36 to 45.00] | 23 [17.16 to 51.54]
  Week 13, improvement: number analyzed (Participants) | 71 | 72
  Week 13, improvement | 35 [31.03 to 67.75] | 20 [14.12 to 47.36]
  Week 13, significant improvement: number analyzed (Participants) | 71 | 72
  Week 13, significant improvement | 11 [6.07 to 34.23] | 5 [1.77 to 23.59]
  Week 25, evident aggravation: number analyzed (Participants) | 70 | 70
  Week 25, evident aggravation | 0 [0.00 to 13.33] | 1 [0.11 to 16.01]
  Week 25, aggravation: number analyzed (Participants) | 70 | 70
  Week 25, aggravation | 1 [0.11 to 16.01] | 1 [0.11 to 16.01]
  Week 25, without changes: number analyzed (Participants) | 70 | 70
  Week 25, without changes | 7 [3.10 to 27.82] | 20 [14.55 to 48.45]
  Week 25, weak improvement: number analyzed (Participants) | 70 | 70
  Week 25, weak improvement | 13 [7.87 to 37.86] | 19 [13.54 to 46.99]
  Week 25, improvement: number analyzed (Participants) | 70 | 70
  Week 25, improvement | 31 [26.69 to 63.44] | 22 [16.62 to 51.31]
  Week 25, significant improvement: number analyzed (Participants) | 70 | 70
  Week 25, significant improvement | 18 [12.54 to 45.52] | 7 [3.10 to 27.82]
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs PLACEBO, ОА Grade II-III; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.005, Chi-squared — The level of significance was set to p <0.05; P-value generated by Chi-squared test was ≤0.005 for each time point

7. Secondary Outcome: Assessment of the Total Number of NSAID Tablets Taken
Description: A patient diary was used to capture data about the number of NSAID Tablets Taken. In case of paracetamol ineffectiveness and pain persistence patient was allowed to take Protocol-permitted NSAID in certain doses.
Time Frame: week 6 (visit 3), week 13 (visit 4), week 25 (visit 5)
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Number; unit: Number of NSAID tablets
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
Number of NSAID tablets | 0 | 0

8. Secondary Outcome: Assessment of the Total Number of Paracetamol Tablets Taken
Description: A patient diary was used to capture data about the number of paracetamol tablets taken.
Time Frame: week 6 (visit 3), week 13 (visit 4), week 25 (visit 5)
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention). The mean number of tablets was calculated taking into account only patients who had received paracetamol.
Measure: Mean (Standard Deviation); unit: mean number of paracetamol taken
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
mean number of paracetamol taken
  Week 6 | 3.08 (3.75) | 6.00 (5.63)
  Week 13 | 1.75 (1.39) | 8.47 (6.67)
  Week 25 | 1.00 (0.00) | 11.79 (9.60)
Statistical Analysis 1: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; The mean number of paracetamol tablets was calculated taking into account only patients who had received paracetamol. ANCOVA was used to detect a difference in means of 2 groups at visit 3 (week 6); Test type: Superiority; p = 0.050, ANCOVA — The threshold for statistical significance was p <0.05
Statistical Analysis 2: Comparison: NOLTREX™, OA Grade II-III vs Placebo, ОА Grade II-III; The mean number of paracetamol tablets was calculated taking into account only patients who had received paracetamol. ANCOVA was used to detect a difference in means of 2 groups at visit 4 (week 13); Test type: Superiority; p = 0.004, ANCOVA — The threshold for statistical significance was p <0.05

9. Secondary Outcome: Patient Exclusion Rates Due to Safety
Description: According to protocol the reasons for withdrawal included health status deterioration, investigator's decision, need in paracetamol use ≥4 days a week during 2 consecutive weeks, individual intolerance or contraindications to the study MD, placebo, paracetamol or any of the protocol-permitted NSAIDs; development of a AE/SAE requiring examination and/or treatment that can significantly affect the study procedures
Time Frame: Week 25
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
participants | 0 [0.00 to 4.99] | 0 [0.00 to 4.99]

10. Secondary Outcome: Exclusion Rate Due to Poor Patient Compliance
Description: According to the protocol the reasons for patients drop-out included major protocol deviations (poor compliance) and withdrawal of informed consent.
Time Frame: Week 25
Population: The intent-to-treat (ITT) population (all randomized patients who received at least one dose of study intervention).
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | NOLTREX™, OA Grade II-III | Placebo, ОА Grade II-III
Number analyzed (Participants) | 72 | 72
participants | 1 [0.04 to 7.50] | 1 [0.04 to 7.50]

ADVERSE EVENTS:
Time Frame: 1 year From 29-Nov-2019 to 17-Nov-2020
Groups:
- NOLTREX™, II-III Grade OA: patients with II-III grade of gonarthrosis will randomised to receive PAHG
  hydrous biopolymer with silver ions "Argiform": 4.0 ml for one injection with one-week interval between injections. Course - 2 injections.
  In NOLTREX™ Group, 5 AEs occurred in 2 (2.78%) patients, and none of them was described as SAE.
- Placebo, II-III Grade ОА: patients with II-III grade of gonarthrosis will randomised to receive saline solution
  saline solution: 4.0 ml for one injection with one-week interval between injections. Course - 2 injections.
  In Placebo Group, 11 AEs occurred in 2 (2.78%) of patients, of them, in 1 (1.39%) patient SAE was registered.
Arm/Group | NOLTREX™, II-III Grade OA | Placebo, II-III Grade ОА
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 1/72
Other Adverse Events (participants affected / at risk) | 5/72 | 11/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOLTREX™, II-III Grade OA (N=72) | Placebo, II-III Grade ОА (N=72)
community-acquired bilateral polysegmental pneumonia caused by coronavirus infection COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Community-acquired bilateral polysegmental pneumonia caused by coronavirus infection COVID-19 (Infections and infestations) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOLTREX™, II-III Grade OA (N=72) | Placebo, II-III Grade ОА (N=72)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Lower back pain
Lumbar spine pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
General weakness. (General disorders) | 1 (1) | 0 (0)
A sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT03897686/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/86/NCT03897686/SAP_001.pdf